CLINICAL TRIAL: NCT03303716
Title: Natural History Study for the ASXL-Related Disorders and Chromatinopathies
Brief Title: ASXL-Related Disorders Natural History Study
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Boston Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Duke University (Other)
Responsible Party: Principal Investigator, Bianca E. Russell, MD, Bianca Russell, MD, University of California, Los Angeles
Other Study IDs: CIN_ASXLHistory_001
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Bohring-Opitz Syndrome; ASXL1 Gene Mutation; Shashi-Pena Syndrome; ASXL2 Gene Mutation; Bainbridge-Ropers Syndrome; ASXL3 Gene Mutation
MeSH Terms: conditions — Bohring syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A registry focused on the natural history, management and treatment of patients with Bohring-Opitz Syndrome (ASXL1), Shashi-Pena Syndrome (ASXL2) and Bainbridge-Ropers Syndrome (ASXL3).

DETAILED DESCRIPTION:
Study participants will be asked to complete a series of brief surveys over time about their medical condition. The researchers will also attain primary medical records.The registry is based at UCLA as the IRB of record with collaborating sites at Boston Children's Hospital, Cincinnati Children's Hospital, and Duke University in a partnership with the Bohring-Opitz Syndrome (BOS) Foundation and ASXL-Rare Research Endowment (ARRE). The BOS Foundation and ARRE are non-profit organizations run by families of patients with ASXL-related disorders that are focused on supporting research. The data is co-managed by the researchers and the family groups. Aggregate data from the Registry will be shared with the participants as well as used for publication. The Registry is HIPPA compliant and follows all the IRB requirements regarding securing and managing patient data.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or molecular diagnosis of an ASXL related disorder

Exclusion Criteria:

* No clinical or molecular diagnosis of an ASXL related disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with molecularly proven or suspected ASXL related disorders
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2037-09 (Estimated); Study Completion 2037-09 (Estimated)

PRIMARY OUTCOMES:
Natural history, treatment and management strategies of ASXL-related disorders | 20 years
  Use participant surveys including the GRDR CDE standard questions to collect data on disease history and management. Attain primary medical records with goal of publications to enhance treatment, management and understanding of the natural history of ASXL gene disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Hann Tan, BMBS, Principal Investigator — Boston Children's Hospital; Loren Pena, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Vandana Shashi, MD, PhD, Principal Investigator — Duke University; Bianca Russell, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided